CLINICAL TRIAL: NCT01659424
Title: Phase II Trial of Preoperative High-dose-rate Endorectal Brachytherapy (BT) FOLFOX Chemotherapy for Stage II/III Rectal Cancer
Brief Title: Phase II Trial of Preoperative High-dose-rate Endorectal Brachytherapy and FOLFOX Chemotherapy for Rectal Cancer
Acronym: HDRBT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Beth Israel Medical Center (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDRBT for Rectal cancer
Record Dates: First submitted 2012-04-24; First posted 2012-08-07 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): This is a single arm study.
  Interventions: Radiation: High Dose Rate Endorectal Brachytherapy (HDR-ERBT)

INTERVENTIONS:
Radiation: High Dose Rate Endorectal Brachytherapy (HDR-ERBT) — Combining pre-operative FOLFOX chemotherapy with HDR-ERBT (Radiation therapy) followed by surgery then additional FOLFOX chemotherapy to decrease the risk of distant metastasis and to maintain excellent locoregional control with decreased morbidity.

SUMMARY:
Standard treatment for rectum cancer is a pre-surgery course of external beam radiotherapy given with chemotherapy at the same time. External beam radiation can increase side effects both short and long-term by exposing normal tissue nearby the tumor such as the bladder, bowel and sexual organs. Instead, this study will use a different way of delivering radiation called brachytherapy to decrease normal tissue radiation exposure. Patient will be given three chemotherapy medications both before and after surgery: oxaliplatin (also called EloxatinTM) in combination with 5-fluorouracil (5-FU) and leucovorin (also called Folinic Acid).

The purpose of this study is to find out whether giving chemotherapy and brachytherapy before surgery can: 1) enable patient's surgeon to successfully remove tumor 2) lower the risk of tumor recurrence 3) avoid patient having the side effects related to chemotherapy and external beam radiation therapy and 4) improve patient's ability to complete chemotherapy.

DETAILED DESCRIPTION:
Summary

Introduction and Rationale:

Over the past 30 years, major advances in adjuvant therapy and surgical techniques have markedly improved cure rates for patients with locoregionally advanced rectal cancer such that pelvic tumor control is over 90%. Preoperative chemoradiation consisting of 5 ½ weeks of external beam radiotherapy combined with radiosensitizing 5-fluorouracil followed by total mesorectal excision (TME) then adjuvant chemotherapy represents the current standard of care. Despite improved survival and locoregional control, disease-free survival have plateaued at rates of 70% because of the high incidence of distant metastasis in about 1/3 of patients.

Clearly, development of more effective systemic therapy approaches to eliminate micrometastatic disease are needed to further improve survival outcomes. The incorporation of oxaliplatin, combined with 5-fluorouracil (FOLFOX), as adjuvant treatment of resected stage II-III colon cancer has led to clinically and statistically significant improvements in disease-free and overall survival in colon cancer. In rectal cancer, FOLFOX has been used primarily after TME but with compliance rates of typically 70%.

One approach to address systemic disease and improve compliance is to treat patients with FOLFOX chemotherapy upfront prior to locoregional therapy. Moreover, incorporating an effective radiation regimen with lower incidence of short and long-term side effects may further enhance compliance to systemic therapy. External beam radiation therapy (EBRT) can increase side effects both acute and chronic toxicity by exposing normal tissue nearby the tumor such as the bladder, bowel, and sexual organs. An appealing technical alternative to EBRT is a brachytherapy (BT) approach using a rectal applicator placed intraluminally in direct contact with the tumor to deliver radiation while sparing adjacent normal organs and decreasing exposure to the pelvic bone marrow. A rectal brachytherapy approach treating over 300 patients has been reported by the McGill group showing equivalent pelvic control, higher pathologic complete response rates and lower short and long-term toxicity. The rectal brachytherapy regimen consists of 4 daily treatments over one week given without chemotherapy which significantly shortens treatment time and cost compared to a standard course of fractionated external beam pelvic radiotherapy. One concern of the rectal brachytherapy approach is that pelvic nodes typically covered in the external beam technique may result in suboptimal outcomes. However, careful patterns of failure studies from a large Dutch preoperative external beam randomized study have shown very low rates of isolated pelvic nodal relapse and minimal benefit of external beam radiotherapy to decrease such failure.

Proposal investigator propose combining pre-operative FOLFOX chemotherapy with high dose rate endorectal brachytherapy followed by surgery and then additional FOLFOX chemotherapy to further improve compliance.

Primary Endpoint The purpose of this study is to find out whether giving chemotherapy and a new technique for delivering radiation therapy before surgery can improve compliance to systemic therapy by 10% from a baseline of 70%.

Secondary Endpoints

1. Locoregional failure
2. Distant Metastasis
3. Bladder, Bowel, Sexual function and Bone Marrow Toxicity
4. Quality of Life
5. Pathologic complete response rates
6. Molecular changes on pre- and post-treatment tumor specimens

Study Design The treatment regimen would consist of 6 cycles of FOLFOX and HDR-ERBT (4 consecutive daily treatments to deliver 26Gy) followed in 6-8 weeks by TME surgery then an additional 6 cycles of FOLFOX chemotherapy after recovery from surgery. HDR-ERBT will be given after 4 cycles of FOLFOX.

*Brachytherapy will be given to subjects at Beth Israel Medical Center only.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the rectum
* T2/3 tumors at ≤ 12cm from the A-V margin (below the peritoneal reflection)
* Tumors with a lumen to allow the positioning of the rectal applicator.
* Tumor of less than 3.5cm thickness documented at the CT Simulator
* Patient should be a suitable candidate for surgery and chemotherapy
* ECOG/WHO performance status 0-1
* Age 18 or older
* No previous history of pelvic radiation or chemotherapy
* Adequate marrow reserve, with absolute neutrophil count greater than or equal to 1.5 x 109/L and platelets greater than or equal to 100 x 109/L.
* Serum creatinine <= 1.5 x ULN; bilirubin <= 1.5 x ULN; ALT<= 2.5 x ULN
* Non pregnant, non-lactating females under active contraception
* No peripheral neuropathy > grade 2

Exclusion Criteria:

* Evidence of necrotic pelvic nodes or ≥ 1 cm
* Evidence of distant metastasis
* Previous pelvic radiation
* Other cancer except for non-melanomatous carcinoma of the skin or CIS of the cervix.
* Presence of multiples small bowel loops trapped within the immediate tumor bed (post hysterectomy or prostatectomy).
* Use of any investigational agent within the 4 weeks preceding enrolment
* Exposure to chemotherapy during the neoadjuvant phase
* Documented distant metastases
* Significant neuropathy
* History of allergic reactions to platin compounds or 5-FU or leucovorin
* Uncontrolled intercurrent illness such as active infection, congestive heart failure or coronary artery disease.
* Psychiatric illness that would limit compliance with study requirements
* Pregnancy or lactation
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Phase II Trial of Preoperative High-dose-rate Endorectal Brachytherapy (BT) Improve Compliance | five years
  Investigator propose combining pre-operative FOLFOX chemotherapy with high dose rate endorectal brachytherapy followed by surgery and then additional FOLFOX chemotherapy to further improve compliance.

SECONDARY OUTCOMES:
Locoregional failure | 5 years
Distant Metastasis | 5 years
Toxicity | 1 year
  Number of participant with Bladder, Bowel, Sexual function and Bone Marrow Toxicity.
4) Quality of Life | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hu, MD, Principal Investigator — Beth Israel Medical Center NY
Locations (2):
- United States (2):
  - Beth Isael Medical Center, New York, New York
  - St-Lukes Roosevelt Hospital Medical Center, New York, New York